CLINICAL TRIAL: NCT00198016
Title: Coil Embolization of Coronary Artery Fistulas: A Single Centre Experience
Brief Title: Coil Embolization of Coronary Artery Fistulas
Status: Completed | Type: Observational
Sponsor: HOSPITEN (Other)
Other Study IDs: HOSPITEN
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2005-08

CONDITIONS: C14; C14907933; C14907933125; G09330582163324; C14280647250
Keywords: coronary fistulas.; coils embolization.

INTERVENTIONS:
Device: Coil

SUMMARY:
Background and Purpose: Congenital coronary artery fistula (CAF) is an uncommon anomaly. In some patients they can became symptomatic, associated with significant morbidity and mortality. We report our experience in percutaneous treatment of CAF.

DETAILED DESCRIPTION:
Congenital coronary artery fistula (CAF) can be defined as a direct communication of a coronary artery with a cardiac chamber, great vessel, or other vascular structure, bypassing the myocardial capillary bed.

CAF is an uncommon anomaly, occurring as an incidental finding in 0.1% to 0.2% of coronary angiograms. They are not gender specific. Many patients have symptoms like congestive heart failure, infective endocarditis, myocardial ischemia, or rupture of an aneurismal fistula. Surgical closure of coronary artery fistula was initially reported in 1983 with low rates of morbidity and mortality.

Percutaneous treatment appeared as an alternative to surgery. Transcatheter closure of CAF was first utilized in 1983. Along this years, with experience and improvements in catheterization equipment and occlusion devices, CAF occlusion have been successfully performed using microcoils.

We report our experience in using microcoils to percutaneous treatment of coronary fistulas.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery fistulas
* Clinical diagnosis of angina, myocardial infarction, left ventricular insufficiency, ventricular enlargement

Exclusion Criteria:

* Age <18 or > 85 years
* Cardiogenic shock _ severe ventricular enlargement

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Zuheir Kabbani, Cardiology, Study Director — HOSPITEN
Locations (1):
- HOSPITEN, Santa Cruz, Tenerife, Spain